CLINICAL TRIAL: NCT05604261
Title: A Multicenter, Randomized, Double-blind, Double-dummy, Positive Drug Parallel Controlled Phase II Clinical Trial to Evaluate Efficacy and Safety of Anaprazole Sodium Enteric-coated Tablets in the Treatment of Reflux Esophagitis
Brief Title: A Study of Anaprazole Sodium Enteric-coated Tablets in the Treatment of Reflux Esophagitis
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Xuanzhu Biopharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 3571-RE-2001
Record Dates: First submitted 2022-10-26; First posted 2022-11-03 (Actual); Last update posted 2022-11-03 (Actual); Status verified 2022-10

CONDITIONS: Reflux Esophagitis; Gastroesophageal Reflux; Esophagitis; Esophageal Motility Disorders; Deglutition Disorders; Esophageal Diseases; Gastrointestinal Diseases
Keywords: Anti-Ulcer Agents; Gastrointestinal Agents; Proton Pump Inhibitors; Enzyme Inhibitors
MeSH Terms: conditions — Esophagitis, Peptic; Gastroesophageal Reflux; Esophagitis; Esophageal Motility Disorders; Deglutition Disorders; Esophageal Diseases; Gastrointestinal Diseases | interventions — Rabeprazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Anaprazole sodium 40 mg QD (Experimental)
  Interventions: Drug: Anaprazole sodium 40 mg
- Anaprazole sodium 60 mg QD (Experimental)
  Interventions: Drug: Anaprazole sodium 60 mg
- Rabeprazole sodium 20 mg QD (Active Comparator)
  Interventions: Drug: Rabeprazole sodium 20 mg

INTERVENTIONS:
Drug: Anaprazole sodium 40 mg — Anaprazole sodium 2 tablets (20 mg/tablet) + Anaprazole sodium dummy tablets 1 tablet (20 mg/tablet) + Rabeprazole sodium dummy tablets 2 tablets (10 mg/tablet) orally once daily within 30-60 minutes before breakfast for 8 weeks (after 4 weeks of continuous treatment, if endoscopy shows reflux esophagitis is cured, treatment is discontinued, into the safety follow-up period).
  Arms: Anaprazole sodium 40 mg QD
Drug: Anaprazole sodium 60 mg — Anaprazole sodium 3 tablets (20 mg/tablet) + Rabeprazole sodium dummy tablets 2 tablets (10 mg/tablet) orally once daily within 30-60 minutes before breakfast for 8 weeks (after 4 weeks of continuous treatment, if endoscopy shows reflux esophagitis is cured, treatment is discontinued, into the safety follow-up period).
  Arms: Anaprazole sodium 60 mg QD
Drug: Rabeprazole sodium 20 mg — Anaprazole sodium dummy tablets 3 tablets (20 mg/tablet) + Rabeprazole sodium 2 tablets (10 mg/tablet) orally once daily within 30-60 minutes before breakfast for 8 weeks (after 4 weeks of continuous treatment, if endoscopy shows reflux esophagitis is cured, treatment is discontinued, into the safety follow-up period).
  Arms: Rabeprazole sodium 20 mg QD

SUMMARY:
A phase 2, randomized, double-blind, double-dummy, positive drug parallel controlled, multicenter trial to evaluate efficacy and safety of within 8 weeks (including 8 weeks) treatment of Anaprazole 40mg QD, 60mg QD compared with Rabeprazole 20mg QD in patients with reflux esophagitis.

DETAILED DESCRIPTION:
This is a multicenter, randomized, double-blind, double-dummy, active drug-parallel-controlled, phase 2 clinical study to evaluate the efficacy and safety of Anaprazole Sodium 40 mg QD and 60 mg QD versus Rabeprazole Sodium 20 mg QD in the treatment of reflux esophagitis in Chinese subjects with reflux esophagitis. The target population for this study was subjects with endoscopically confirmed reflux esophagitis. All potential participants will provide informed consent, and those who provide informed consent will enter the Screening Period (Day -7 to Day -1) and be assessed for screening eligibility according to the inclusion and exclusion criteria. The study is expected to enroll approximately 156 subjects with reflux esophagitis (LA classification grades A-D) who meet enrollment criteria (and none of the exclusion criteria), and eligible subjects will be randomized into 3 groups (Anaprazole Sodium 40 mg QD, 60 mg QD, and Rabeprazole Sodium 20 mg QD) in a 1:1: 1 ratio according to a predefined randomization table, with 52 subjects in each group. All subjects take the corresponding study drug within 30-60 minutes before breakfast for 4 or 8 consecutive weeks (subjects were followed up at Week 4 of treatment, and if the subject'endoscopy indicated that the reflux esophagitis was healed, the healed subject ended study treatment and entered safety follow-up. Subjects who were not cured were to continue treatment until 8 weeks if endoscopy at 4 weeks of treatment indicated that reflux esophagitis was not cured.). All subjects complete treatment at 4 or 8 weeks of treatment and were followed for safety. At the end of the study, statistical analysis will be performed on the efficacy and safety indicators of the study drug to compare the efficacy and safety of Anaprazole sodium and rabeprazole sodium in the treatment of reflux esophagitis. Participants will primarily be assessed for the cure rate of reflux esophagitis based on endoscopy of 3 groups. Participants' safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects clearly understand and voluntarily participate in this study, sign the informed consent form and voluntarily comply with the study procedures;
2. Age ≥ 18 years and ≤ 70 years, male or female;
3. Endoscopic diagnosis of reflux esophagitis (LA classification criteria grades A-D) within 7 days prior to randomization.

Exclusion Criteria:

Subjects who meet any of the following criteria will not be allowed to participate in this study:

Past medical history

1. Subjects whose primary diseases that are not suitable for participating in the clinical trial cannot be effectively controlled in the investigator 's opinion, such as patients with previous severe heart, brain, lung, liver, kidney and other systemic diseases;
2. Patients with previous concomitant diseases that may affect esophageal motility or motility, which may still affect the efficacy evaluation (e.g., eosinophilic esophagitis, esophageal varices, scleroderma, viral infection or fungal infection, esophageal stenosis, etc.) at the investigator 's discretion, or with a history of esophageal radiotherapy or esophageal cryotherapy;
3. History of previous surgical procedures that could affect the esophagus (eg, fundoplication and mechanical dilatation for esophageal strictures), or history of gastric or duodenal surgery, excluding endoscopic removal of benign polyps;
4. Subjects with active peptic ulcer, active upper/lower gastrointestinal bleeding confirmed by esophagogastroduodenoscopy (EGD) within 30 days prior to randomization;
5. Subjects with previous Zollinger-Ellison syndrome, achalasia, secondary esophageal motility disorder, irritable bowel syndrome, inflammatory bowel disease;
6. Prior malignancy or treatment for malignancy within 5 years prior to randomization (except cured cutaneous basal cell carcinoma or cervical carcinoma in situ);
7. Subjects who have a previous history of psychiatric disorders (except for patients with current psychiatric disorders who are stable and not under medication control as judged by the investigator), or a history of drug or alcohol abuse within 12 months prior to Screening.

   General/Laboratory Tests
8. Abnormal liver function at screening: aspartate aminotransferase (AST) and/or alanine aminotransferase (ALT) ≥ 1.5 × ULN and/or total bilirubin (TBIL) ≥ 1.5 × ULN;
9. Abnormal renal function at screening: serum creatinine (Cr) ≥ 1.2 × ULN/blood urea nitrogen (BU)/blood urea nitrogen (BUN) ≥ 1.2 × ULN; Other conditions
10. Patients unable to undergo esophagogastroduodenoscopy (EGD);
11. Patients who are allergic to Annarazole Sodium or Rabeprazole Sodium and other drug ingredients or components that may be used in the study;
12. Use of therapeutic doses of drugs for gastroesophageal reflux disease such as proton pump inhibitors, potassium-competitive acid blockers, histamine H2 receptor antagonists, mucosal protective drugs, prokinetic drugs, anti-Helicobacter pylori drugs, and Chinese patent medicines for gastroesophageal reflux disease within 7 days before randomization;
13. Subjects who may affect the efficacy and safety evaluation due to alcohol, drug and drug withdrawal during the study;
14. Pregnant or lactating women, subjects with fertility plan from 30 days before randomization to half a year after the end of the trial;
15. Participation in another drug clinical trial (defined as receiving investigational product or placebo) within 3 months prior to randomization;
16. Other conditions that the investigator considers the subject unsuitable for this clinical trial.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 156 (Estimated)
Dates: Start 2022-12 (Estimated); Primary Completion 2023-07 (Estimated); Study Completion 2024-03 (Estimated)

PRIMARY OUTCOMES:
The endoscopic healing rate of reflux esophagitis within 8 weeks (including 8 weeks) | Treatment of 4 weeks or 8 weeks
  The endoscopic ulcer healing rate is defined as the percentage of patients with reflux esophagitis healed evaluated by blinded independency central reading. Reflux esophagitis is evaluated by endoscopy as per LA Classification.

SECONDARY OUTCOMES:
The rate of improvement in each individual symptom (daytime reflux) | Treatment of 4 weeks or 8 weeks
  The assessment of improvement of daytime reflux is evaluated in terms of severity and frequency. Mean severity scores are calculated for the first 7 days of the 4-week and 8-week visits, respectively. Mean score = sum of individual scores recorded over 7 days/number of days recorded.
  Complete response: mean score/score reduced to 0. Improvement:mean score/score reduced to 1. Ineffective: no change or increase in mean score/score. Complete response rate = number of complete response cases/total number of cases × 100%. Improvement rate = number of improved cases/total number of cases × 100%.
The rate of improvement in each individual symptom (daytime heartburn) | Treatment of 4 weeks or 8 weeks
  The assessment of improvement of daytime heartburn is evaluated in terms of severity and frequency. Mean severity scores are calculated for the first 7 days of the 4-week and 8-week visits, respectively. Mean score = sum of individual scores recorded over 7 days/number of days recorded.
  Complete response: mean score/score reduced to 0. Improvement:mean score/score reduced to 1. Ineffective: no change or increase in mean score/score. Complete response rate = number of complete response cases/total number of cases × 100%. Improvement rate = number of improved cases/total number of cases × 100%.
The rate of improvement in each individual symptom (nighttime reflux) | Treatment of 4 weeks or 8 weeks
  The assessment of improvement of nighttime reflux is evaluated in terms of severity and frequency. Mean severity scores are calculated for the first 7 days of the 4-week and 8-week visits, respectively. Mean score = sum of individual scores recorded over 7 days/number of days recorded.
  Complete response: mean score/score reduced to 0. Improvement:mean score/score reduced to 1. Ineffective: no change or increase in mean score/score. Complete response rate = number of complete response cases/total number of cases × 100%. Improvement rate = number of improved cases/total number of cases × 100%.
The rate of improvement in each individual symptom (nighttime heartburn) | Treatment of 4 weeks or 8 weeks
  The assessment of improvement of nighttime heartburn is evaluated in terms of severity and frequency of each of the four individual symptoms. Mean severity scores are calculated for the first 7 days of the 4-week and 8-week visits, respectively. Mean score = sum of individual scores recorded over 7 days/number of days recorded.
  Complete response: mean score/score reduced to 0. Improvement:mean score/score reduced to 1. Ineffective: no change or increase in mean score/score. Complete response rate = number of complete response cases/total number of cases × 100%. Improvement rate = number of improved cases/total number of cases × 100%.
Change From Baseline in gastroesophageal reflux disease health-related quality of life scale (GERD-HRQL) score | Treatment of 4 weeks or 8 weeks
  GERD related quality of life (QoL) is assessed with the "gastroesophageal reflux disease - health related quality of life" (GERD-HRQL) questionnaire. QoL is measured at baseline and at six months after treatment. The scale contains 10 questions and a symptom control satisfaction survey, which focuses on heartburn, acid reflux, swallowing function, and drug efficacy. Each question is scored according to a scoring criteria of 6 scores (0 indicates no symptoms, 5 indicates intolerable symptoms, and affects daily activities), and the total score is the sum of the scores of each item (0-50 points in total), with higher scores indicating worse quality of life. Satisfaction is divided into three levels: dissatisfaction, moderate, and satisfaction. Change in GERD-HRQL score = total GERD-HRQL score after treatment - total GERD-HRQL score before treatment.
Adverse events | Through study completion, an average of 1 year
  Number of participants with treatment-related adverse events as assessed by CTCAE v5.0.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Changhai Hospital, Shanghai, Shanghai Municipality, China